CLINICAL TRIAL: NCT05872815
Title: Precision Drug Use of Immunosuppressants Guided by Population Pharmacokinetics/Pharmacodynamic Models in Kidney Transplant Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-50
Record Dates: First submitted 2023-04-19; First posted 2023-05-24 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Kidney Transplantation; Immunosuppressive Agents
Keywords: Population pharmacokinetics/pharmacodynamics; Immunosuppressive Agents; Kidney transplantation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. Construct a population pharmacokinetic/pharmacodynamic model of tacrolimus in kidney transplant patients, and explore the quantitative relationship between combination drugs and gene polymorphisms on the safety and efficacy of tacrolimus in kidney transplant patients;
2. Based on the established pharmacokinetic/pharmacodynamic model of tacrolimus population in kidney transplant patients, combined with combined drugs, gene polymorphisms and other factors for simulation, predict the steady-state trough concentration and efficacy of tacrolimus in kidney transplant patients taking triple drugs (tacrolimus, mycophenolate mofetil/mycophenol sodium enteric-coated tablets, glucocorticoids), and apply the model to the real world to explore the optimal initial dose and maintenance therapeutic dose of tacrolimus, so as to achieve individualized and precise treatment and guide the rational clinical use of drugs.
3. Clarify the value of precision medicine guided by population pharmacokinetics/pharmacodynamics models in clinical practice.

DETAILED DESCRIPTION:
This is a retrospective study. It is proposed to combine the classical basic principles of pharmacokinetics with mathematical statistical models, and use nonlinear mixed effect model (NONMEM) or other population pharmacokinetics/pharmacodynamics software to establish a population pharmacokinetic/pharmacodynamic model of tacrolimus in kidney transplant patients, and elucidate the combination of drugs, demographic factors, pathophysiological factors, genotype, The quantitative effect of comorbid diseases and drugs on the steady-state trough concentration and efficacy of tacrolimus in kidney transplant patients, so as to realize individualized and precise treatment of kidney transplant patients through model simulation and prediction of steady-state trough concentration and efficacy after taking drugs.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing kidney transplantation for the first time.
* Anti-rejection therapy with triple immunosuppressant (tacrolimus + mycophenolate mofetil + glucocorticoids).

Exclusion Criteria:

* The patient's medication status is unclear and there is a lack of relevant results of laboratory test indicators.
* The patient has undergone multi-organ or combined liver and kidney transplantation or has a history of liver and kidney transplantation.
* Transplantation failure or death.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All of the included population was kidney transplant patients,and all of they used triple immunosuppressant (tacrolimus + mycophenolate mofetil + glucocorticoids) for anti-rejection therapy,the results of laboratory could be collected.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Drug plasma tough concentrations | Blood samples were collected 30minutes before administration
  The tough concentrations of tacrolimus are as regard as the PK parameters
Immune factors levels(CD4+、CD8+、CD4+/CD8+、CD4+%、CD8+%) | The Immune factors levels were collected 30minutes before administration
  The Immune factors levels are as regard as the PD parameters

SECONDARY OUTCOMES:
Clinical indicators | Follow-up after kidney transplantation was 6 months
  Incidence of acute rejection,Incidence of tacrolimus adverse reactions and other advers are as regard as the PD parameters

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Chongqing Medical University, Chongqing, China